CLINICAL TRIAL: NCT06942078
Title: Cryoneurolysis as an Interim Pain Control Strategy in Patients Awaiting Total Hip and Knee Arthroplasty: a Prospective Observational Study
Brief Title: Cryoneurolysis in Patients Awaiting Total Hip and Knee Arthroplasty
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Calgary (Other)
Responsible Party: Principal Investigator, Ryan Endersby, Clinical Assistant Professor, Department of Anesthesiology, Perioperative and Pain Medicine, University of Calgary
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: REB25-0319
Record Dates: First submitted 2025-04-16; First posted 2025-04-24 (Actual); Last update posted 2025-09-25 (Actual); Status verified 2025-09

CONDITIONS: Hip Arthropathy; Knee Arthropathy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Cryoneurolysis (Experimental): Participants will receive a diagnostic nerve block with local anesthetic. This block will be performed on nerves that supply the hip joint or knee joint depending on location of osteoarthritis. If pain relief is greater than 50%, cryoneurolysis will be performed targeting nerves that supply the hip or knee joint with very low temperatures.
  Interventions: Procedure: Cryoneurolysis

INTERVENTIONS:
Procedure: Cryoneurolysis — Targeting of specific nerves related to surgical procedure using very low temperatures

SUMMARY:
During the COVID-19 pandemic, there was a drastic increase in surgical wait times across Canada, notably for patients awaiting total knee and hip arthroplasty. Currently the average wait time for total hip arthroplasty (THA) in Alberta is 16 weeks with the 90th percentile of wait times being 47 weeks. The average wait for total knee arthroplasty (TKA) in Alberta is 20 weeks with the 90th percentile of wait times being 60 weeks. As the waitlist for these surgeries grows and with limited resources to increase the number of surgeries being performed, there is a critical need for strategies to manage the pain experienced by patients during these long waiting periods.

Many patients awaiting surgery are placed onto long-term opioid therapy to manage their pain. There are, however, significant risks associated with the extended use of opioids for pain management, such as addiction, opioid abuse, increased risk of overdose, increased risk of fractures, and increased risk of adverse cardiac events. Recognizing these risks, different strategies need to be employed to attempt to minimize the opioid burden faced by those waiting for surgery. One potential strategy is to utilize regional anesthesia for analgesia rather than relying on opioids. Regional anesthesia with nerve blocks using local anesthetic has been used in the management of preoperative pain for patients awaiting surgery for hip fracture and has been shown to be effective in reducing pain, opioid use, and the risk of serious adverse effects. However, for patients with hip fractures, their surgery usually occurs within 36 hours due to significant risks which occur beyond that timeframe. For patients waiting for THA and TKA, the surgical wait time could be weeks to months. Providing daily nerve blocks or even weekly catheters for an individual waiting up to a year for surgery is not sustainable and carries significant risks with repeated injections. New regional anesthesia techniques lasting a longer period of time are needed.

One promising intervention is to utilize cryoneurolysis. Cryoneurolysis involves treating targeted nerves using extremely low temperatures. This disrupts nerve conduction and pain impulses. Importantly, connective tissue components of the nerve are left intact allowing for regeneration over time. Because of this, cryoneurolysis is a well-established treatment for chronic and acute pain due to its effectiveness and low risk safety profile. While cryoneurolysis is well-established in its use treating chronic and surgical pain, one limitation is that it is focused primarily on postoperative pain. Our study intends to primarily evaluate the efficacy of cryoneurolysis as a preoperative pain management intervention. Establishing the use of cryoneurolysis for preoperative pain will provide a valuable resource for reducing the pain patients experience while awaiting surgery, leading to decreased opioid use and improved overall well-being. The investigators will be recruiting 30 participants total (15 having TKA and 15 having THA) that will be given cryoneurolysis while waiting for their surgery.

ELIGIBILITY:
Inclusion Criteria:

* Currently awaiting THA or TKA (have signed consent for surgery)
* Osteoarthritis as a primary diagnosis for THA or TKA
* Currently taking regular daily opioids for at least one month
* No allergies to local aesthetics
* Speaks and understands English
* Over 18 years old
* Lives within a 1-hour distance of the hospital where the study is taking place or willing to travel to the hospital for the interventions and follow up.

Exclusion Criteria:

* If surgery is expected to be completed within 1 month of the intervention as this would limit our ability to evaluate the effectiveness of the cryoneurolysis procedure
* Allergies to local anesthetics
* Inability to communicate with investigators
* Opioid use disorder
* History of severe psychiatric or medical conditions which hinder effective communication
* Living more than 1 hour away from the hospital where the study is taking place or unable to travel to the hospital for the interventions and follow up
* Body mass Index (BMI) ≥40
* Any contraindications specific to percutaneous cryoneurolysis such as history of bleeding diathesis, any active infections at the procedural site, cold urticaria, cryofibrinogenemia, cryoglobulinemia, paroxysmal cold hemoglobinuria, or Raynaud's disease (see Ilfeld & Finneran, 2020)
* Use of therapeutic anticoagulation
* Diagnosis of Non-Osteoarthritis as the cause for THA or TKA
* Other chronic pain condition which patients may be taking opioids to control the pain (e.g. Fibromyalgia or Complex Regional Pain Syndrome)
* Less than 50% reduction in pain with diagnostic blocks using 0.5% bupivacaine

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-10-01 (Estimated); Primary Completion 2027-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Oral Morphine Equivalent Consumption | Pre-intervention, 2-weeks, 4-weeks, 8-weeks, 6 months, and 1-year post-intervention; 2-weeks, 6-weeks, 12-weeks postoperative
  Daily Oral Morphine Equivalent Consumption

SECONDARY OUTCOMES:
NRS Pain Score | Pre-intervention, 2-weeks, 4-weeks, 8-weeks, 6 months, and 1-year post-intervention; 2-weeks, 6-weeks, 12-weeks postoperative
  Numerical Rating Scale Pain Score
EQ-5D Score | Pre-intervention, 2-weeks, 4-weeks, 8-weeks, 6 months, and 1-year post-intervention; 2-weeks, 6-weeks, 12-weeks postoperative
  EuroQol 5-Dimension Score
WOMAC Score | Pre-intervention, 2-weeks, 4-weeks, 8-weeks, 6 months, and 1-year post-intervention; 2-weeks, 6-weeks, 12-weeks postoperative
  Western Ontario and McMaster Universities Osteoarthritis Index Score

CONTACTS AND LOCATIONS:
Overall Officials: Ryan Endersby, MD, Principal Investigator — University of Calgary

IPD SHARING:
Plan to Share IPD: No